CLINICAL TRIAL: NCT00529100
Title: A Phase I/II Study of Concurrent Pemetrexed/Cisplatin/Radiation in Stage IIIA/B Non-Small Cell Lung Cancer
Brief Title: Concurrent Pemetrexed, Cisplatin and Radiation Therapy in Patients With Stage IIIA/B Non Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10259; H3E-CA-JMHU (Other: Eli Lilly and Company); NCT00470730 (obsolete NCT alias)
Record Dates: First submitted 2007-09-12; First posted 2007-09-14 (Estimated); Results first posted 2011-09-28 (Estimated); Last update posted 2013-07-09 (Estimated); Status verified 2013-07

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pemetrexed/Cisplatin/Radiation Phase 1 (Experimental): Treatment included: radiation as 61-65 Gray (Gy) in 33-35 fractions if 2-phase treatment and 62-66 Gy in 31-33 fractions if 1-phase treatment; concurrent pemetrexed intravenous (IV) bolus with doses escalating from 300 milligrams per square meter (mg/m^2) IV through 500 mg/m^2 IV on Days 1 and 22; concurrent cisplatin 25 mg/m^2 IV on Days 1-3 and 22-24 for Cohorts 1-3 and cisplatin 20 mg/m^2 IV on Days 1-5 and 22-26 for Cohort 4. Participants then received 2 additional consolidation cycles repeated every 3 weeks (q3 weeks) of pemetrexed 500 mg/m^2 IV and cisplatin 75 mg/m^2 IV.
  Interventions: Drug: Pemetrexed Phase 1; Drug: Cisplatin Phase 1; Procedure: Radiation Therapy
- Pemetrexed/Cisplatin/Radiation Phase 2 (Experimental): Treatment included: radiation, 61-65 Gy in 33-35 fractions if 2-phase treatment and 62-66 Gy in 31-33 fractions if 1-phase treatment; concurrent phase pemetrexed IV bolus as determined by Phase 1 trial to be 500 mg/m^2 IV on Days 1 and 22 ; concurrent cisplatin 20 mg/m^2 IV as determined by Phase 1 trial with cycles commencing on Days 1 and 22; 2 additional consolidation cycles (q3 weeks) of pemetrexed 500 mg/m^2 IV and cisplatin 75 mg/m^2 IV.
  Interventions: Procedure: Radiation Therapy; Drug: Pemetrexed Phase 2; Drug: Cisplatin Phase 2

INTERVENTIONS:
Drug: Pemetrexed Phase 1 — 300 mg/m^2 IV, Days 1 and 22; intermediate dose escalation level of 400 mg/m^2 IV; then 500 mg/m^2 IV, repeated every 21 days (q 21 days) x 2 cycles
  Other Names: LY231514; Alimta
  Arms: Pemetrexed/Cisplatin/Radiation Phase 1
Drug: Cisplatin Phase 1 — Cohorts 1-3: 25 mg/m^2 IV, Days 1-3 and 22-24 then 75 mg/m^2 IV, q21 days x 2 cycles
  Cohort 4 carried into Phase 2: 20 mg/m^2 IV, Days 1-5 and 22-26 then 75 mg/m^2 IV, q21 days x 2 cycles.
  Arms: Pemetrexed/Cisplatin/Radiation Phase 1
Procedure: Radiation Therapy — Phases 1 and 2: 61-65 Gy in 33-35 fractions
Drug: Pemetrexed Phase 2 — Concurrent phase pemetrexed IV bolus as determined by Phase 1 trial to be 500 mg/m^2 IV on Days 1 and 22.
  Other Names: LY231514; Alimta
  Arms: Pemetrexed/Cisplatin/Radiation Phase 2
Drug: Cisplatin Phase 2 — Phase 2 (Cohort 4 carried over from Phase 1): 20 mg/m^2 IV, Days 1-5 and 22-26 then 75 mg/m^2 IV, q21 days x 2 cycles.
  Arms: Pemetrexed/Cisplatin/Radiation Phase 2

SUMMARY:
Measure the 1 year survival of non small cell lung cancer (NSCLC) patients who are being treated with pemetrexed in combination with cisplatin and radiation.

ELIGIBILITY:
Inclusion Criteria:

Some of the requirements to be in this study are:

* Patient must be at least 18 years old.
* Patient must have been diagnosed with non-small cell lung cancer.
* Patient must be able to visit the doctor's office once a week.
* Patient must have adequate blood, liver, lungs and kidney function within the requirements of this study.
* Female patients of child-bearing potential must test negative for pregnancy at the time of enrollment based on a serum pregnancy test. Male and female patients must agree to use a reliable method of birth control during and for 3 months following the last dose of study drug.

Exclusion Criteria:

Patients cannot participate in this study for any of the following reasons:

* Patient has previously had chemotherapy.
* Patient has previously had thoracic radiation therapy.
* Patient has received treatment within the last 30 days with a drug that has not received approval by Health Canada for any indication at the time of study entry.
* Female patient is pregnant or breast-feeding.
* Patient is unsuitable to participate in the study in the opinion of the investigator.
* Patient is unable or unwilling to take folic acid, vitamin B12 supplementation, or dexamethasone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2005-12; Primary Completion 2010-08 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern time (UTC/GMT- 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- Canada (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edmonton, Alberta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamilton, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ottawa, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toronto, Ontario

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 16 participants entered Phase 1 of the study. A total of 39 participants were analyzed in Phase 2, which included data from 6 Phase 1 participants.
Groups:
- Pemetrexed/Cisplatin/Radiation Phase 1: Treatment included: radiation as 61-65 Gray (Gy) in 33-35 fractions if 2-phase treatment and 62-66 Gy in 31-33 fractions if 1-phase treatment; concurrent pemetrexed intravenous (IV) bolus with doses escalating from 300 milligrams per square meter (mg/m^2) IV through 500 mg/m^2 IV on Days 1 and 22; concurrent cisplatin 25 mg/m^2 IV on Days 1-3 and 22-24 for the first three cohorts and cisplatin 20 mg/m^2 IV on Days 1-5 and 22-26 for Cohort 4. Participants then received 2 additional consolidation cycles (every 3 weeks [q3 weeks]) of pemetrexed 500 mg/m^2 IV and cisplatin 75 mg/m^2 IV.
- Pemetrexed/Cisplatin/Radiation Phase 2: Treatment included: radiation, 61-65 Gy in 33-35 fractions if 2-phase treatment and 62-66 Gy in 31-33 fractions if 1-phase treatment; concurrent pemetrexed IV bolus as determined by Phase 1 trial on Days 1 and 22; concurrent cisplatin as determined by Phase 1 trial with cycles commencing on Days 1 and 22; and 2 additional consolidation cycles (q3 weeks) of pemetrexed 500 mg/m^2 IV and cisplatin 75 mg/m^2 IV.
Period: Overall Study
Arm/Group | Pemetrexed/Cisplatin/Radiation Phase 1 | Pemetrexed/Cisplatin/Radiation Phase 2
Started | 16 | 33
Received at Least 1 Dose of Study Drug | 16 | 33
Completed | 16 | 24
Not Completed | 0 | 9
Not completed — Adverse Event | 0 | 5
Not completed — Protocol Violation | 0 | 1
Not completed — Progressive Disease | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Participant Ineligibility | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received study drug in Phase 1, Phase 1 and 2, or Phase 2.
Groups:
- Pemetrexed/Cisplatin/Radiation Phase 1: Participants were strictly in Phase 1. Treatment included: radiation as 61-65 Gray (Gy) in 33-35 fractions if 2-phase treatment and 62-66 Gy in 31-33 fractions if 1-phase treatment; concurrent pemetrexed intravenous (IV) bolus with doses escalating from 300 milligrams per square meter (mg/m^2) IV through 500 mg/m^2 on Days 1 and 22; concurrent cisplatin 25 mg/m^2 IV on Days 1-3 and 22-24 for the first three cohorts and cisplatin 20 mg/m^2 IV on Days 1-5 and 22-26 for Cohort 4. Participants then received 2 additional consolidation cycles (q3 weeks) of pemetrexed 500 mg/m^2 IV and cisplatin 75 mg/m^2 IV.
- Pemetrexed/Cisplatin/Radiation Phase 1-Phase 2: Participants were overlap in Phase 1 and Phase 2.
- Pemetrexed/Cisplatin/Radiation Phase 2: Participants were strictly in Phase 2. Treatment included: radiation, 61-65 Gy in 33-35 fractions if 2-phase treatment and 62-66 Gy in 31-33 fractions if 1-phase treatment; concurrent pemetrexed IV bolus as determined by Phase 1 trial on Days 1 and 22; concurrent cisplatin as determined by Phase 1 trial with cycles commencing on Days 1 and 22; 2 additional consolidation cycles (q3 weeks) of pemetrexed 500 mg/m^2 IV and cisplatin 75 mg/m2 IV.
- Total: Total of all reporting groups
Arm/Group | Pemetrexed/Cisplatin/Radiation Phase 1 | Pemetrexed/Cisplatin/Radiation Phase 1-Phase 2 | Pemetrexed/Cisplatin/Radiation Phase 2 | Total
Number analyzed (Participants) | 10 | 6 | 33 | 49
Age Continuous [Mean (Standard Deviation); unit: years] | 60.3 (8.0) | 64.3 (8.1) | 61.2 (10.5) | 61.4 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 18 | 27
  Male | 4 | 3 | 15 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 6 | 30 | 46
  Unknown or Not Reported | 0 | 0 | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 2
  White | 9 | 5 | 27 | 41
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 10 | 6 | 33 | 49

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Maximum Tolerated Dose (MTD) of Pemetrexed in Combination With Cisplatin and Radiation Therapy
Description: Recommended Phase 2 MTD was highest dose at which no more than 1 of 6 participants experienced dose level toxicity (DLT). DLT=(1) Grade 3/4 dysphagia/esophagitis, leukopenia, thrombocytopenia, febrile neutropenia, fatigue/malaise, pneumonitis, dermatitis, persistent elevation of bilirubin/alkaline phosphatase/aspartate aminotransferase only if resulting in delay of radiotherapy >1 week, delay of pemetrexed/cisplatin Cycle 2 >2 weeks, or delay of pemetrexed/cisplatin Cycle 3 past 5 weeks after radiotherapy; (2) other Grade 3 or 4 toxicity possibly related to concurrent treatment administration.
Time Frame: Baseline to measured progressive disease (PD; up to 1 year)
Population: The treated population included all participants who received at least 1 dose of either study therapy (that is, pemetrexed, cisplatin, or radiation).
Measure: Number; unit: milligrams per square meter (mg/m^2)
Groups:
- Pemetrexed/Cisplatin/Radiation Phase 1: Treatment included: radiation as 61-65 Gray (Gy) in 33-35 fractions if two-phase treatment and 62-66 Gy in 31-33 fractions if one-phase treatment; concurrent pemetrexed intravenous (IV) bolus with doses escalating from 300 milligrams per square meter (mg/m^2) through 500 mg/m^2 on Days 1 and 22; concurrent cisplatin 25 mg/m^2 on Days 1-3 and 22-24 for the first three cohorts and cisplatin 20 mg/m^2 on days 1-5 and 22-26 for cohort four. Participants then received two additional consolidation cycles (q3 weekly) of pemetrexed 500 mg/m^2 and cisplatin 75 mg/m^2.
Arm/Group | Pemetrexed/Cisplatin/Radiation Phase 1
Number analyzed (Participants) | 16
milligrams per square meter (mg/m^2)
  Concurrent Phase MTD: Pemetrexed | 500
  Concurrent Phase MTD: Cisplatin | 20
  Consolidation Phase MTD: Pemetrexed | 500
  Consolidation Phase MTD: Cisplatin | 75

2. Primary Outcome: Phase 2: Percentage of Participants With Overall Survival (OS) at 1 Year
Description: OS was defined as the time from date of enrollment to death due to any cause.
Time Frame: Baseline to date of death from any cause (up to 1 year)
Population: The treated population was considered the primary analysis population for the efficacy endpoints. The efficacy analysis was also completed on the protocol-qualified (PQ)population to assess the sensitivity of the results.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Pemetrexed/Cisplatin/Radiation Phase 2: Treatment included: radiation, 61-65 Gy in 33-35 fractions if two-phase treatment and 62-66 Gy in 31-33 fractions if one-phase treatment; concurrent pemetrexed 500 mg/m^2 as determined by phase 1 trial on Days 1 and 22; concurrent cisplatin 20 mg/m^2 as determined by phase 1 trial with cycles commencing on Days 1 and 22; two additional consolidation cycles (q3 weekly) of pemetrexed 500 mg/m^2 and cisplatin 75 mg/m2.
Arm/Group | Pemetrexed/Cisplatin/Radiation Phase 2
Number analyzed (Participants) | 39
percentage of participants | 79.0 [66.1 to 92.0]

3. Secondary Outcome: Phase 1: Number of Participants With Adverse Events (AE; Toxicity)
Description: A listing of AEs is located in the Reported Adverse Event module.
Time Frame: Baseline to measured PD (up to 1 year)
Population: The treated population was used for this analysis and included all participants who received at least 1 dose of either study therapy (pemetrexed, cisplatin, or radiation).
Measure: Number; unit: participants
Groups:
- Pemetrexed/Cisplatin/Radiation Phase 1: Treatment included: radiation as 61-65 Gray (Gy) in 33-35 fractions if two-phase treatment and 62-66 Gy in 31-33 fractions if one-phase treatment; concurrent pemetrexed intravenous (IV) bolus with doses escalating from 300 milligrams per square meter (mg/m^2) through 500 mg/m^2 on Days 1 and 22; concurrent cisplatin 25 mg/m^2 on Days 1-3 and 22-24 for the first three cohorts and cisplatin 20 mg/m^2 on Days 1-5 and 22-26 for Cohort 4. Participants then received two additional consolidation cycles (q3 weekly) of pemetrexed 500 mg/m^2 and cisplatin 75 mg/m^2.
Arm/Group | Pemetrexed/Cisplatin/Radiation Phase 1
Number analyzed (Participants) | 10
participants
  Serious Adverse Events (SAEs) | 5
  Other Non-serious Adverse Events (AEs) | 10

4. Secondary Outcome: Phase 2: Percentage of Participants With Overall Survival (OS) at 2 Years and 3 Years
Description: OS was defined as the time from date of enrollment to death due to any cause.
Time Frame: Baseline and 2 years and 3 years
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Pemetrexed/Cisplatin/Radiation Phase 2: Treatment included: radiation, 61-65 Gy in 33-35 fractions if two-phase treatment and 62-66 Gy in 31-33 fractions if one-phase treatment; concurrent pemetrexed IV bolus as determined by Phase 1 trial on Days 1 and 22; concurrent cisplatin as determined by Phase 1 trial with cycles commencing on Days 1 and 22; and two additional consolidation cycles (q3 weeks) of pemetrexed 500 mg/m^2 and cisplatin 75 mg/m^2.
Arm/Group | Pemetrexed/Cisplatin/Radiation Phase 2
Number analyzed (Participants) | 39
percentage of participants
  2 years | 56.4 [40.8 to 72.0]
  3 years | 46.2 [30.5 to 61.8]

5. Secondary Outcome: Phase 2: Time to Progressive Disease (PD)
Description: Time to PD was defined as the time from study enrollment to the first date of objective disease progression as defined by Response Evaluation Criteria in Solid Tumors (RECIST 1.0) as at least a 20% increase in the sum of the longest diameter (LD) of target lesions as references the smallest sum LD recorded since treatment started or the appearance of 1 or more new lesions. Time to PD was censored at the date of death if death was due to other cause. For participants not known to have died as of the data cut-off date and who did not have PD, time to PD was censored at the last progression-free disease assessment. For participants who received subsequent cancer therapy (after discontinuation from the study therapy) before PD, time to PD was censored at the date of subsequent cancer therapy initiation.
Time Frame: Baseline to measured PD (up to 3 years)
Population: The treated population was used for this analysis and included all participants who received at least 1 dose of either study therapy (pemetrexed, cisplatin, or radiation). Eleven participants were censored.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed/Cisplatin/Radiation Phase 2
Number analyzed (Participants) | 39
months | 13.7 [10.2 to 19.2]

6. Secondary Outcome: Phase 2: Percentage of Participants With Progression Free Survival (PFS)
Description: The percentage of participants not known to have died as of the data cut-off date or last contact and who did not have PD.
Time Frame: Baseline and 1 year and 2 years and 3 years
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemetrexed/Cisplatin/Radiation Phase 2
Number analyzed (Participants) | 39
percentage of participants
  1 Year | 48.7 [33.0 to 64.4]
  2 Years | 30.8 [16.3 to 45.3]
  3 Years | 20.2 [7.5 to 32.9]

7. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the period from study entry until PD, death, or date of last contact. For participants not known to have died as of the data cut-off date and who did not have PD, the PFS date was censored at the last contact date (contacts considered in the determination of last progression free disease assessment).
Time Frame: Baseline to measured PD (up to 36 months)
Population: The treated population was used for this analysis and included all participants who received at least 1 dose of either study therapy (pemetrexed, cisplatin, or radiation). Eight participants were censored.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed/Cisplatin/Radiation Phase 2
Number analyzed (Participants) | 39
months | 11.8 [9.8 to 19.2]

8. Secondary Outcome: Phase 2: Percentage of Participants With Objective Tumor Response (Response Rate)
Description: Response using Response Evaluation Criteria In Solid Tumors (RECIST 1.0). Complete Response (CR)=disappearance of all target lesions; Partial Response (PR)=30% decrease in sum of longest diameter of target lesions; Progressive Disease (PD)=20% increase in sum of longest diameter of target lesions; Stable Disease (SD)=small changes that do not meet above criteria. Objective response rate (%)=number of objective responders divided by the number of participants with measurable disease * 100, where objective responders are those participants who have met criteria either for CR or PR.
Time Frame: Baseline to measured PD (up to 3 years)
Population: The treated population was used for this analysis and included all participants who received at least 1 dose of either study therapy (pemetrexed, cisplatin, or radiation) and with measurable disease.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemetrexed/Cisplatin/Radiation Phase 2
Number analyzed (Participants) | 37
percentage of participants
  Complete Response | 0 [0 to 0]
  Partial Response | 45.95 [29.89 to 62.00]

9. Secondary Outcome: Phase 2: Site of Progressive Disease (PD)
Description: Summarized participants with local (progression within the sites of initial disease)/regional (disease progression adjacent to but not within the site of initial disease at the start of treatment), distant (disease progression that is blood borne to other parts of the body, including outside the chest or involving the contralateral lung), and local + distant sites of disease. Objective PD is defined by Response Evaluation Criteria in Solid Tumors (RECIST 1.0) as at least a 20% increase in the sum of the longest diameter (LD) of target lesions as references the smallest sum LD recorded since treatment started or the appearance of 1 or more new lesions.
Time Frame: Baseline to measured PD (up to 3 years)
Population: The treated population was used for this analysis and included all participants who received at least 1 dose of either study therapy (pemetrexed, cisplatin, or radiation) and who had PD.
Measure: Number; unit: participants
Arm/Group | Pemetrexed/Cisplatin/Radiation Phase 2
Number analyzed (Participants) | 27
participants
  Local/Regional | 8
  Distant | 17
  Local + Distant | 1
  Unknown | 1

ADVERSE EVENTS:
Time Frame: Serious Adverse Events (SAE) and other Non-Serious Adverse Events were collected during study treatment only, participants received study drug for 4 cycles of 21 days per cycle.
Groups:
- Pemetrexed/Cisplatin/Radiation Phase 1: Treatment included: radiation as 61-65 Gray (Gy) in 33-35 fractions if two-phase treatment and 62-66 Gy in 31-33 fractions if one-phase treatment; concurrent pemetrexed intravenous (IV) bolus with doses escalating from 300 milligrams per square meter (mg/m^2) through 500 mg/m^2 on Days 1 and 22; concurrent cisplatin 25 mg/m^2 on Days 1-3 and 22-24 for the first three cohorts and cisplatin 20 mg/m^2 on Days 1-5 and 22-26 for Cohort 4. Participants then received two additional consolidation cycles (q3 weeks) of pemetrexed 500 mg/m^2 and cisplatin 75 mg/m^2.
- Pemetrexed/Cisplatin/Radiation Phase 1-2: Cohort 4 data from Phase (Ph) 1 was included in the Ph 2 analysis as Cohort 4 was the established dose from Ph 1.
  Ph 1: radiation as 61-65 Gray (Gy) in 33-35 fractions if 2-phase treatment/62-66 Gy in 31-33 fractions if 1-phase treatment; concurrent pemetrexed IV bolus with doses escalating from 300 milligrams per square meter (mg/m^2) through 500 mg/m^2 on Days 1 and 22; concurrent cisplatin 25 mg/m^2 on Days 1-3 and 22-24 for the first 3 cohorts and cisplatin 20 mg/m^2 on Days 1-5 and 22-26 for Cohort 4. Participants then received 2 additional consolidation cycles (q3 weeks) of pemetrexed 500 mg/m^2 and cisplatin 75 mg/m^2.
  Ph 2: radiation, 61-65 Gy in 33-35 fractions if 2-phase treatment/62-66 Gy in 31-33 fractions if 1-phase treatment; concurrent pemetrexed IV bolus from Ph 1 trial on Days 1 and 22; concurrent cisplatin from Ph 1 trial with cycles commencing on Days 1 and 22; and 2 additional consolidation cycles (q3 weeks) of pemetrexed 500 mg/m^2 and cisplatin 75 mg/m^2.
Arm/Group | Pemetrexed/Cisplatin/Radiation Phase 1 | Pemetrexed/Cisplatin/Radiation Phase 1-2 | Pemetrexed/Cisplatin/Radiation Phase 2
Serious Adverse Events (participants affected / at risk) | 5/10 | 0/6 | 9/33
Other Adverse Events (participants affected / at risk) | 10/10 | 6/6 | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed/Cisplatin/Radiation Phase 1 (N=10) | Pemetrexed/Cisplatin/Radiation Phase 1-2 (N=6) | Pemetrexed/Cisplatin/Radiation Phase 2 (N=33)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Fatigue (General disorders) | 0 (0) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 2 (2) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed/Cisplatin/Radiation Phase 1 (N=10) | Pemetrexed/Cisplatin/Radiation Phase 1-2 (N=6) | Pemetrexed/Cisplatin/Radiation Phase 2 (N=33)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 6 (22) | 28 (96)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 3 (5)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (4) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 2 (8) | 1 (2)
Dry eye (Eye disorders) | 0 (0) | 1 (4) | 0 (0)
Keratoconjunctivitis sicca (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 2 (8) | 1 (4)
Photophobia (Eye disorders) | 0 (0) | 2 (5) | 0 (0)
Vision blurred (Eye disorders) | 1 (2) | 1 (1) | 2 (2)
Vitreous floaters (Eye disorders) | 0 (0) | 1 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (4) | 0 (0) | 4 (4)
Constipation (Gastrointestinal disorders) | 8 (19) | 5 (7) | 18 (34)
Diarrhoea (Gastrointestinal disorders) | 5 (10) | 2 (3) | 11 (16)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 4 (11) | 1 (2) | 10 (27)
Dysphagia (Gastrointestinal disorders) | 5 (17) | 2 (8) | 15 (38)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (6)
Nausea (Gastrointestinal disorders) | 6 (14) | 2 (7) | 28 (67)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 2 (5) | 11 (24)
Oesophageal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oesophageal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3)
Oesophageal stenosis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 5 (11) | 3 (9) | 20 (48)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (2) | 5 (6)
Vomiting (Gastrointestinal disorders) | 6 (11) | 1 (2) | 20 (34)
Chest pain (General disorders) | 3 (9) | 0 (0) | 9 (17)
Chills (General disorders) | 1 (3) | 0 (0) | 1 (1)
Fatigue (General disorders) | 9 (28) | 6 (16) | 30 (87)
General symptom (General disorders) | 1 (1) | 0 (0) | 0 (0)
Ill-defined disorder (General disorders) | 1 (4) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 1 (2) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 4 (10) | 2 (5) | 6 (12)
Pain (General disorders) | 4 (11) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 3 (3)
Sensation of foreign body (General disorders) | 0 (0) | 0 (0) | 2 (6)
Unevaluable event (General disorders) | 1 (1) | 0 (0) | 0 (0)
Immune system disorder (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 2 (4)
Opportunistic infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Radiation skin injury (Injury, poisoning and procedural complications) | 1 (1) | 5 (10) | 18 (41)
Activated partial thromboplastin time prolonged (Investigations) | 2 (3) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (5) | 0 (0) | 6 (9)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 1 (1) | 8 (9)
Blood albumin decreased (Investigations) | 6 (8) | 0 (0) | 5 (13)
Blood alkaline phosphatase increased (Investigations) | 2 (4) | 1 (2) | 3 (9)
Blood bicarbonate (Investigations) | 0 (0) | 2 (2) | 1 (1)
Blood bicarbonate decreased (Investigations) | 0 (0) | 0 (0) | 2 (4)
Blood bilirubin increased (Investigations) | 2 (2) | 0 (0) | 1 (1)
Blood calcium decreased (Investigations) | 4 (8) | 0 (0) | 0 (0)
Blood calcium increased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 3 (10) | 0 (0) | 8 (16)
Blood glucose increased (Investigations) | 9 (26) | 0 (0) | 0 (0)
Blood magnesium decreased (Investigations) | 5 (15) | 0 (0) | 4 (9)
Blood phosphorus decreased (Investigations) | 4 (7) | 0 (0) | 2 (3)
Blood potassium decreased (Investigations) | 1 (3) | 0 (0) | 0 (0)
Blood potassium increased (Investigations) | 2 (6) | 0 (0) | 0 (0)
Blood sodium decreased (Investigations) | 5 (10) | 0 (0) | 0 (0)
Blood sodium increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 2 (3)
Ear, nose and throat examination abnormal (Investigations) | 1 (4) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 9 (32) | 5 (18) | 26 (79)
International normalised ratio increased (Investigations) | 1 (2) | 0 (0) | 3 (5)
Lymphocyte count decreased (Investigations) | 10 (36) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 9 (28) | 6 (19) | 24 (56)
Platelet count decreased (Investigations) | 8 (21) | 6 (10) | 16 (29)
Weight decreased (Investigations) | 4 (9) | 0 (0) | 6 (10)
White blood cell count decreased (Investigations) | 9 (32) | 6 (19) | 27 (77)
Decreased appetite (Metabolism and nutrition disorders) | 5 (12) | 2 (3) | 17 (43)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 8 (9)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (9) | 24 (53)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 8 (15)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (4)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (7) | 8 (19)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (5) | 12 (16)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 9 (12)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (9) | 14 (32)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 3 (6) | 24 (40)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 6 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (8) | 1 (3) | 3 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (6) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (8)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (5) | 1 (1) | 1 (2)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 3 (6) | 2 (2) | 9 (17)
Dysgeusia (Nervous system disorders) | 0 (0) | 2 (4) | 3 (8)
Headache (Nervous system disorders) | 2 (5) | 2 (6) | 5 (6)
Peripheral motor neuropathy (Nervous system disorders) | 1 (4) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (14) | 1 (2) | 5 (10)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 4 (4)
Anxiety (Psychiatric disorders) | 4 (10) | 0 (0) | 5 (10)
Depression (Psychiatric disorders) | 2 (8) | 0 (0) | 1 (3)
Insomnia (Psychiatric disorders) | 2 (6) | 2 (3) | 4 (7)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (29) | 2 (2) | 15 (31)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 (12) | 0 (0) | 7 (14)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (23) | 0 (0) | 7 (14)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 1 (4) | 8 (14)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 1 (4) | 4 (6)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (7) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (4)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 2 (8) | 0 (0) | 0 (0)
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (4) | 1 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (16)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 (5) | 0 (0) | 0 (0)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 5 (14) | 0 (0) | 1 (6)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (4) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (3) | 1 (1) | 4 (8)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (6) | 7 (17)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 5 (14)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Hot flush (Vascular disorders) | 1 (2) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (6) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 4 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less